CLINICAL TRIAL: NCT03155464
Title: A Prospective Study of the Utility of Intraoperative, Quantitative Indocyanine Green Angiography in Microvascular Surgery for Systemic Scerlosis
Brief Title: Intraoperative ICG for Systemic Sclerosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The device that was going to be studied was removed by Duke University shortly after the study was approved.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00078686
Record Dates: First submitted 2017-04-24; First posted 2017-05-16 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Systemic Sclerosis
Keywords: indocyanine-green; systemic scerlosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: This study will enroll participants in a 1:1 randomized study design. Participants will serve as their own controls. A consecutive series of patients will be randomized to either Group 1 or 2. Randomization will occur through 40 sealed, opaque sequentially numbered envelopes containing the randomization. Those that qualify and sign consent will be randomized 24hrs prior to surgery. The randomization envelopes will be stored in a locked filing cabinet within the clinical research coordinators office. The subject will know what treatment arm they are in prior to surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Other): Order of two elements of surgical procedure: patients in group 1 will receive sympathectomy prior to bypass during the surgical procedure.
  Indocyanine Green (ICG) will be used in both groups.
  Interventions: Procedure: Order of two elements of surgical procedure; Drug: Indocyanine Green
- Group 2 (Other): Order of two elements of surgical procedure: Patients in group 2 will receive bypass prior to sympathectomy during the surgical procedure.
  Indocyanine Green (ICG) will be used in both groups.
  Interventions: Procedure: Order of two elements of surgical procedure; Drug: Indocyanine Green

INTERVENTIONS:
Procedure: Order of two elements of surgical procedure — Please see the arm/group descriptions for the order of elements of the surgical procedure in group 1 and group 2.
Drug: Indocyanine Green — Intraoperative ICG has been validated to correlate to postoperative outcomes. ICG is administered by means of peripheral or central intravenous access, is excreted exclusively by the liver into the bile, and is not associated with risk for nephrotoxicity. We will be using a concentration of 2.5mg/cc. 12.5mg will be administered at each injection of ICG. Complete washout of the ICG occurs after 15 minutes, plenty of time considering the interval surgery that must occur. As per the protocol, ICG will be administered 3 times during the surgery. The patients will receive a total of 37.5mg of ICG, well below the recommended threshold of 2mg/kg. No significant toxic effects have been observed in humans with the high dose of 5 mg/kg of body weight.
  Other Names: ICG

SUMMARY:
The primary objective of this study is to evaluate the relative intraoperative improvement in perfusion between arterial reconstruction and sympathectomies with quantitative ICG. A minimum of 40 patients, 20 Sympathectomy Prior to Bypass (group 1) and 20 Bypass Prior to Sympathectomy (group 2), will be recruited for this study. This study will enroll participants in a one to one randomized study design. There is the potential risk of loss of confidentiality. The study involves the intraoperative assessment of perfusion by quantitative ICG. ICG is FDA approved for this usage and will be used according to its labeling. Assessment involves intraoperative quantitative ICG data, questionnaires, and patient and physician assessments. There are no additional physical risks associated with participating in this study over and above that of the planned arterial reconstruction (bypass) and sympathectomies.The information collected will be kept confidential and will comply with the HIPAA.

DETAILED DESCRIPTION:
A minimum of 40 patients, 20 Sympathectomy Prior to Bypass (group 1) and 20 Bypass Prior to Sympathectomy (group 2), will be recruited for this study. This study will enroll participants in a 1:1 randomized study design. Participants will serve as their own controls. A consecutive series of patients will be randomized to either Group 1 or 2. Randomization will occur through 40 sealed, opaque sequentially numbered envelopes containing the randomization. Those that qualify and sign consent will be randomized 24hrs prior to surgery. The randomization envelopes will be stored in a locked filing cabinet within the clinical research coordinators office. The subject will know what treatment arm they are in prior to surgery.

Patients will be randomized to Group 1 or 2. If patients are randomized to Group 1, patients will receive sympathectomy prior to bypass during the surgical procedure (see below). If patients are randomized to Group 2, they will received bypass prior to sympathectomy during the surgical procedure (see below). Patients in both groups will be in the study for the next 12 months. Normal clinical practice will not change. Patients in both groups will be examined before surgery. If they provide consent to participate, demographical data, comorbidities, the number and severity of digital ulcerations, and baseline outcome measures for the Michigan Hand Outcome Questionnaire, Disabilities of the Arm, Shoulder and Hand and the Visual Analogue Scale for Pain will be collected.

Patients in both groups will return to the office for routine follow-up at 2 weeks for wound care. The next study visit will occur at 6 weeks. At that time, outcome measures will be again administered and data collected. In accordance with standard clinical practice, the patients will return to the office for examination again at 6 months and 1 year. At these times, the primary clinical outcomes will be collected as well as the patient reported outcomes.

These are normal visits, not outside the scope of routine clinical practice. Intraoperative ICG is also within the scope of routine clinical practice. The dose of ICG and the number of times that it is administered to subjects is the same as in standard of care.

ICG is administered by means of peripheral or central intravenous access, is excreted exclusively by the liver into the bile, and is not associated with risk for nephrotoxicity. The laser diode array utilized by the SPY System emits a near-infrared wavelength that does not require the use of protective eyewear or other safety equipment. The investigators will be using a concentration of 2.5mg/cc. 12.5mg will be administered at each injection of ICG. Complete washout of the ICG occurs after 15 minutes, plenty of time considering the interval surgery that must occur. As per the protocol, ICG will be administered 3 times during the surgery. The patients will receive a total of 37.5mg of ICG, well below the recommended threshold of 2mg/kg. Of note, No significant toxic effects have been observed in humans with the high dose of 5 mg/kg of body weight.

ELIGIBILITY:
Inclusion Criteria:

* o Patient has signed an IRB approved, study specific Informed Patient Consent Form.

  * Patient is a male or non-pregnant female age 18 - 85 years at time of study enrollment.
  * Patient has a diagnosis of a systemic sclerosis with vascular obstruction of the hand resulting in digital ischemia, ulceration, and/or gangrene and have failed nonoperative treatments.
  * Patient is willing and able to comply with postoperative scheduled clinical evaluations.

Exclusion Criteria:

* • Patient is undergoing revision surgery.

  • Patient has a diagnosis of avascular necrosis or inflammatory arthritis.
* If, during surgery, the arterial reconstruction could not be performed because the vessel was damaged to the point where there was no appropriate site for a bypass anastomosis.

  * Patient is a prisoner
  * Pregnant women confirmed by testing prior to surgery, and nursing mothers
  * Patient has an allergy to iodine confirmed during initial history and on day of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Change in perfusion | Baseline-One Year Follow-up
  To compare the relative intraoperative change in perfusion between arterial reconstruction and sympathectomies with quantitative ICG.

SECONDARY OUTCOMES:
Intraoperative change in hand and digit perfusion | Baseline-One Year Follow-up
  To document the immediate intraoperative quantitative change in hand and digit perfusion in combined arterial reconstruction and sympathectomies in patients with systemic sclerosis using intraoperative quantitative ICG.

OTHER OUTCOMES:
Comparison of clinical and intraoperative quantitative ICG measurements | Baseline-One Year Follow-up
  Correlation of primary clinical measures with results of intraoperative quantitative ICG at 1 year postoperative
Change in Michigan Hand Outcome Questionnaire | Baseline-One Year Follow-up
  Change in Michigan Hand Outcome Questionnaire
Change in Visual Analogue Scale for Pain (VAS) | Baseline-One Year Follow-up
  Change in Visual Analogue Scale for Pain (VAS); patient reported level of pain which is then measured (distance from 0 in mm)
Change in Disability of the Arm, Shoulder, and Hand Questionnaire (DASH) | Baseline-One Year Follow-up
  Change in DASH score; scale of 0-100. 30 questions in total with optional work and optional sports/activities questions (with 4 questions each)
Complete healing of all ulcers | 1 Year Follow-up
  Complete healing of all ulcers (yes/no)
Number of all ulcers | 1 Year Follow-up
  Number of all ulcers
Need for amputation by the end of one-year follow-up | 1-year follow-up
  Need for amputation by the end of one-year follow-up (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Mithani, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No